CLINICAL TRIAL: NCT03783429
Title: Digoxin Evaluation in Chronic Heart Failure: Investigational Study In Outpatients in the Netherlands
Acronym: DECISION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Disphar International B.V. (Industry); Teva Nederland BV (Unknown); Tiofarma BV (Unknown); Netherlands Heart Foundation (Other); Werkgroep Cardiologische centra Nederland (Unknown)
Responsible Party: Principal Investigator, M. Rienstra, Prof. Dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DECISION trial
Record Dates: First submitted 2018-12-13; First posted 2018-12-21 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Digoxin; Atrial fibrillation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Digoxin

STUDY DESIGN:
Intervention Model Description: A national, multicenter, randomized, double-blind placebo controlled, clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group will receive low-dose digoxin
  Interventions: Drug: Digoxin
- Placebo group (Placebo Comparator): The placebo group will receive a matching placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Digoxin — Digoxin tablets will be given orally
  Arms: Intervention group
Drug: Placebos — Placebo tablets will be given orally
  Arms: Placebo group

SUMMARY:
Digoxin is the oldest, market-authorized drug for heart failure (HF), and very cheap. A large trial with digoxin, the DIG trial, executed in the early nineties revealed a highly significant reduction in HF hospitalizations, but no effect on mortality. A post-hoc analysis of the DIG trial suggests that low serum concentrations of digoxin may not only improve HF hospitalizations but also mortality in chronic HF patients. To confirm these retrospective analyses, a prospective, randomized, placebo-controlled trial is necessary to establish the position of digoxin in the contemporary treatment of HF. Therefore, the investigators examine whether low-level, aiming for serum concentrations 0.5-0.9ng/mL, digoxin is beneficial in HF patients with reduced or mid-range ejection fractions (LVEF <50%).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18year
2. Outpatients with chronic HF, New York Heart Association [NYHA] class II - ambulatory IV
3. LVEF<50%
4. Serum NT-proBNP concentrations:

   Previous HF hospitalization ≤ 1 year before randomisation ≥400pg/mL if sinus rhythm; ≥800pg/mL if AF Previous HF hospitalization > 1 year before randomisation or in the absence of HF hospitalizations ≥ 600pg/mL if sinus rhythm; ≥1000 pg/mL if AF

   BNP concentrations:

   Previous HF hospitalization ≤ 1 year before randomisation ≥100pg/mL if sinus rhythm; ≥200pg/mL if AF Previous HF hospitalization > 1 year before randomisation or in absence of HF hospitalization ≥150pg/mL if sinus rhythm; ≥250pg/mL if AF.
5. ≥14 days stable on guideline-recommended therapy (doses and number of therapies as tolerated by each patient)

Exclusion Criteria:

1. Heart rate ≤60bpm (if sinus rhythm); heart rate ≤70bpm (if AF)
2. History of HF hospitalization ≤7days
3. History of myocardial infarction, myocarditis, percutaneous intervention, RCT, pacemaker/ICD implantation, cardiac surgery or stroke ≤30 days
4. Estimated glomerular filtration rate (eGFR), ≤30ml/min/1.73m2
5. The presence of a mechanical assist device
6. Use of inotropic drugs (dopamine, dobutamine, (nor)adrenaline, and milrinon)
7. Scheduled for mechanical assist device or heart transplant
8. Other non-cardiac conditions with limited life expectancy (≤ duration of the study)
9. Amyloid, hypertrophic obstructive or constrictive cardiomyopathy
10. Accessory atrio-ventricular pathway (e.g. Wolf-Parkinson-White syndrome)
11. (Intermittent) complete heart block or second-degree AV block type Mobitz without pace maker or ICD
12. Severe (grade III/III) aortic valve disease
13. Complex congenital heart disease
14. Proven hypersensitivity to digoxin (prior side effects)
15. Concomitant medication that interacts with digoxin
16. Use of digoxin ≤6 months prior to inclusion
17. Participation in another (intervention) clinical trial (registry studies not included)
18. Women who are pregnant, breastfeeding or may be considering pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Composite of repeated HF hospitalizations, urgent HF Visits, and cardiovascular death | Median of 3 years

SECONDARY OUTCOMES:
All-cause mortality | Median of 3 years
Cardiovascular death | Median of 3 years
(Repeated) HF hospitalization | Median of 3 years
Cost-effectiveness assessed by the Medical Consumption Questionnaire | Median of 3 years
Urgent HF hospital visits | Median of 3 years

OTHER OUTCOMES:
All-cause hospitalizations | Median of 3 years
Unscheduled cardiovascular hospital visits | Median of 3 years
Days alive out of hospital | Median of 3 years
Quality of Life assessed by the EUROQOL-5D-5L questionnaire | Median of 3 years
  Quality of Life is assessed by questions about mobility, selfcare, daily activity, pain and anxiety. The questions about mobility, selfcare and daily activity range from 'no problem doing activity' to 'not able to do activity'. The questions about pain and anxiety range from 'not at all present' to 'extremely present'.
  The last question in the questionnaire asks how a person rates his or her health in the present day, ranging from 0-100, where 0 is the worst health imaginable, and 100 is the best health imaginable.
Heart rate in both AF and sinus rhythm | Median of 3 years
To assess side effects (SUSARs) associated with study medication | Median of 3 years
Initiation of (recurrence of) AF in patients with sinus rhythm at baseline | Median of 3 years
Conversion to sinus rhythm and maintenance of sinus rhythm in patients with AF at baseline | Median of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Rienstra, MD, PhD, Principal Investigator — University Medical Center Groningen; Peter van der Meer, MD, PhD, Principal Investigator — University Medical Center Groningen; Dirk J van Veldhuisen, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (44):
- Netherlands (44):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Zorggroep Twente, Almelo
  - Meander Medisch Centrum, Amersfoort
  - BovenIJ Ziekenhuis, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooi, Blaricum
  - Amphia Ziekenhuis, Breda
  - Ijsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Van Weel Bethesda, Dirksland
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Scheper Ziekenhuis, Emmen
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Beatrix Ziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - University Medical Center Groningen, Groningen
  - Spaarne Gasthuis, Haarlem
  - Saxenburgh MC, Hardenberg
  - Ziekenhuis St Jansdal, Harderwijk
  - Zuyderland Medisch Centrum, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Bethesda, Hoogeveen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis, Leiden
  - Maastricht UMC+, Maastricht
  - Isala Diaconessenhuis, Meppel
  - Radboud University Medical Center, Nijmegen
  - Bravis ziekenhuis, Roosendaal
  - Erasmus Medisch Centrum, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Franciscus Vlietland, Schiedam
  - Antonius Ziekenhuis Sneek, Sneek
  - Refaja, Stadskanaal
  - Haaglanden Medisch Centrum, The Hague
  - Elisabeth-Tweesteden Ziekenhuis, Tilburg
  - Diak. Utrecht, Utrecht
  - Máxima Medisch Centrum, Veldhoven
  - Zaans Medisch Centrum, Zaandam

REFERENCES:
- [Derived] van Veldhuisen DJ, Rienstra M, Mosterd A, Alings AM, van Asselt ADJ, Bouvy ML, Tijssen JGP, Schaap J, van der Wall EE, Voors AA, Boorsma EM, Lok DJA, Crijns HJGM, Schut A, Vijver MAT, Voordes GHD, de Vos AH, Maas-Soer EL, Smit NW, Touw DJ, Samuel M, van der Meer P; DECISION Investigators and Committees. Efficacy and safety of low-dose digoxin in patients with heart failure. Rationale and design of the DECISION trial. Eur J Heart Fail. 2024 Oct;26(10):2223-2230. doi: 10.1002/ejhf.3428. Epub 2024 Aug 30. PMID 39212246